CLINICAL TRIAL: NCT06856850
Title: Disease Biosignatures in ALS/FTD Spectrum: New Impactful Biological Perspectives Beyond Clinical Approaches
Acronym: SPECTRALS
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: PNRR MCNT2-2023-12377336
Record Dates: First submitted 2025-02-11; First posted 2025-03-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis); FTD; Neuropathic; Psychiatric Disorders; Idiopathic Intracranial Hypertension; Frontotemporal Dementia (FTD)
Keywords: Amyotrophic lateral sclerosis; frontotemporal dementia; microbiota; miRNA; protein-NMR; TDP-43; endocytic disfunction; seed amplification assay; peripheral biomarker
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Mental Disorders; Pseudotumor Cerebri; Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Diagnosis of ALS/FTD disease spectrum is challenging because it largely relies on clinical symptoms. Identifying novel biomarkers is essential for a paradigm shift towards a more precise biological-based diagnosis. To achieve this aim, having access to proper specimens and analytical methods is crucial. Our team of experts in neurology, biology, chemistry, physics, and AI will explore ALS/FTD from novel perspectives using transcriptomics, proteomics, genomics and other innovative approaches to analyzing easily accessible tissues. The seed amplification assay (SAA) will be also exploited to detect pathological TDP-43. This project aims to create disease fingerprints useful for patient stratification and monitoring of disease progression, and to evaluate the therapeutic efficacy in clinical trials, thus overcoming the limits of clinical interpretation. Discovering new biomarkers and cellular pathways will improve the diagnosis and treatment of these devastating diseases.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) and frontotemporal dementia (FTD) are considered two manifestations of the same disease continuum, sharing common clinical, genetic and pathological features. Both diseases can even co-occur in the same patient, however, the underlying mechanisms triggering ALS, FTD or their mixed phenotype are not fully understood. Unfortunately, reliable biomarkers for ALS/FTD clinical diagnosis are still lacking. The aim of this project is to employ a cutting-edge, multidisciplinary approach to investigate not only traditional cerebrospinal fluid (CSF) samples, but also other easily accessible tissues such as skin, olfactory mucosa (OM), serum and tears. This project intends to uncover new biomarkers able to recognize ALS/FTD clinical phenotypes, strengthen the clinical diagnosis of specific phenotypes (e.g. bulbar vs spinal onset ALS), predict patients at risk of developing a mixed disease phenotype (ALS+FTD or vice versa), evaluate the efficacy of therapeutic treatments and capable to unveiling specific biological mechanisms involved in the onset and progression of each disease. The added value of the project is that it will explore ALS/FTD from a peripheral point of view by using tissues that have yet to be thoroughly examined in this field of research. These tissues will either be subjected to direct analysis for biomarker discovery or processed to perform cell and structural studies useful to deepen our understanding of the ALS/FTD neurodegenerative process and uncover new druggable molecules or mechanisms. To achieve our objectives, the first year of the project will be dedicated to enrolling patients, performing also a retrospective study using already available CSF, serum, tears, and OM samples collected from an extensively characterized cohort of patients with bALS, sALS, FTD as well as subjects with other non-neurodegenerative neurological conditions (NNC). These samples will be subjected to the following analyses (1) NGS, (2) Simoa (to quantify NfL, tau, phospho-tau, and beta-amyloid proteins), (3) Microfluidic (to determine miRNA and long non-coding RNA profiles), (4) Bioplex (to evaluate the innate-adaptive immunity pathway); (5) Seed amplification assay (to detect peripheral pathological TDP-43), and (6) MiSeq Illumina (to analyze microbiota composition). For microfluidic and Bioplex analyses the retrospective study will serve for biomarker discovery. Whereas, for Simoa, SAA and MiSeq analyses this study will allow the collection of pivotal preliminary data and fine-tuning of the analytical procedures. The applicants have already obtained promising data showing that the miRNA profile in serum and TDP-43 content in OM (SAA) could discriminate between bALS and Sals. These findings suggest that molecular and biological profiling is feasible and could tangibly impact the diagnosis of ALS/FTD. The second year of the study will focus on subjecting the newly collected samples to the same analyses as previously described, either for biomarker validation or for collecting all the necessary and essential data to determine whether and to what extent some peripheral alterations actually differ among pathologies. All the data will be processed by the Data Science Center group (expert bioinformaticians, statisticians, mathematicians and neurobiologists) to assess whether our findings allow for the identification of disease biosignatures in ALS/FTD spectrum.

The research group is composed of four operative units (OUs): Fondazione IRCCS Istituto Neurologico Carlo Besta (UO1), Università degli Studi di Napoli "Federico II" (UO2), Consorzio Interuniversitario Risonanze Magnetiche Metallo Proteine (UO3) and Azienda Ospedaliero Universitaria di Sassari (UO4). It has been decided to include a group from Sardinia (UO4) because it is one of the Italian regions with the highest incidence of ALS and will contribute to the enrollment of patients with more heterogeneous clinical presentations. OU1 and UO4 will be responsible for selecting retrospective biological samples and recruiting ALS/FTD and NNC patients in the first year of the study. CSF, blood, tears, skin, and OM samples have been or will be collected using standardized and shared procedures by OU1 and UO4 from a total of sALS (n=105), bALS (n=32), FTD (n=66) and NNC (n=27) patients. A subset of samples collected from sALS (n=45), bALS (n=12), FTD (n=30) and NNC (n=12) patients is already available at UO1 and UO4 and will be analyzed during the first year of new patient enrollment. All recruited subjects will undergo extensive clinical and neuropsychological assessments and will be subjected to the Burghart Sniffin' Sticks test before CSF, blood, OM, skin and tears sampling. Samples will be distributed and analyzed by each UO as follow: CSF will be prepared either for Simoa analysis at UO4 or for (1) miRNA and long non-coding RNA, and (2) SAA analyses at UO1. Blood will be immediately processed at UO1 and UO4 to isolate the serum fraction that will be analyzed at UO4 (Simoa measurement of NfL, amyloid-beta, tau and phosphorylated at threonine 181 tau (p-tau) levels) and UO1 (evaluation of miRNA and long non-coding RNA profiles and evaluation of the innate-adaptive immunity pathway). Tears will be prepared for miRNA and long non-coding RNA or for SAA analyses at UO1. OM will be prepared for (1) miRNA and long non-coding RNA, (2) SAA and (3) microbiota analyses at UO1. Finally, the skin will be prepared for (1) miRNA and long noncoding RNA or (2) SAA analyses at UO1 and will be processed to obtain primary cell fibroblasts that will be sent to UO2 for (3) cell biology studies including super-resolution microscopy analysis of intracellular aggregates and molecular characterization of their internalization/degradation pathways. Finally, UO3 will (1) produce recombinant TDP-43 (for SAA analyses performed at UO1) possessing special features useful to produce NMR spectra of good quality for detailed structural characterization and (2) analyze selected SAA products by protein-NMR. All data generated in this project, including all relevant clinical and psychological information, will be analyzed by members of the Data Science Center (DSC) group that has been recently created at UO1. DSC combines the expertise of bioinformaticians, statisticians, mathematicians and neurobiologists with the aim of applying sophisticated analytical methodologies to clinical, omics, and imaging data. Finally, other collaborators (see appropriate section) working at UO3 will assist with protein-NMR study. Thus, synergistic collaboration among all UOs is vital to achieving the aims of the project.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria for ALS (Brooks et al., 2000; de Carvalho M., 2008), FTD (GornoTempini et al., 2011; Rascovsky et al., 2011)

Exclusion Criteria:

* na

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spinal-ALS (sALS, n=60), Bulbar-ALS (Bals,n=20), FTD (n=36), and NNC (n=10)
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of SAA accuracy in detecting misfolded TDP-43 in CSF, skin, OM, and tears of ALS and FTD patients. | 24 months
  the primary outcome of the study will involve investigating the distribution of misfolded TDP-43, a protein associated with amyotrophic lateral sclerosis (ALS) and frontotemporal dementia (FTD), using ultrasensitive techniques namely Seed Amplification Assays (SAA). These assays will be employed to detect minute amounts of misfolded TDP-43 in cerebrospinal fluid (CSF), olfactory mucosa (OM), serum, skin, and tears from patients, with a clinical diagnosis of bulbar ALS (bALS; n=32), spinal ALS (sALS; n=105), FTD (n=66), and other non-neurodegenerative neurological conditions (NNC; n=27). By analyzing multiple peripheral tissues from the same patients, the generation of a disease biological fingerprint, obtained by integrating SAA analysis, other biochemical tests together with clinical and instrumental findings will be attempted. We aim to explore the reliability of this approach to improve the clinical diagnosis of ALS and FTD by allowing patient stratification.

SECONDARY OUTCOMES:
Diagnostic and prognostic peripheral biomarkers identification through Simoa | 18 months
  To analyze if the levels of total-tau (pg/mL), phosphorylated tau (pg/mL), neurofilament light chains (NfL, pg/mL) and beta-amyloid proteins (pg/mL) are altered in the biological samples analysed (serum and CSF) compared to NNC and if these values differ in such a way that might help us to discriminate the pathologies (sALS, bALS, FTD). The assessment of these components will be pursued using Simoa.
Diagnostic and prognostic peripheral biomarkers identification through Microfluidic analysis | 18 months
  To determine the miRNA and long non-coding RNA profiles of the biological samples analysed (serum, CSF, OM, skin and tears), the TaqManTM Array Human MicroRNA-Card will be used.
  Bioinformatic analysis will be performed using tools and customized pipelines to identify differentially expressed (DE) miRNAs/lncRNAs in ALS and FTD samples compared to NNC. Validation of the top-ranked DE miRNA/lncRNA will be performed. Receiver operating characteristic (ROC) curves and the area under the curve (AUC) will be calculated to assess the ability of each miRNA/lncRNA to differentiate among groups.
Diagnostic and prognostic peripheral biomarkers identification through multiplex immunoassays | 18 months
  To evaluate the innate-adaptive immunity pathway, serum samples will undergo multiplex immunoassays analysis with the Bio-Plex Pro Human Cytokine multiplex kits on the Bioplex 200 system to analyze the levels of molecules, including interleukin (IL)-1ß, IL-4, IL-6, IL-10, IL-17A, IL-17F, IL-21, IL-22, IL-23, IL-31, IL-33 (pg/mL), tumor necrosis factor-alpha (TNF-a; pg/mL), and interferon-gamma (IFN-y; pg/mL)
Metagenomic analysis to evaluate the microbiota composition | 12 months
  CSF and OM will be subjected to metagenomic analysis to evaluate the microbiota composition (eubiosis/dysbiosis), by MiSeq Illumina analysis. Total bacterial DNA will be extracted from CSF and OM samples using the QIAamp DNA Microbiome Kit. The V3-V4 region of the 16S rRNA gene will be amplified using gene-specific primers. 16S libraries will be prepared and completed using the KAPA HiFi HT ReadyMix, following Illumina Nextera DNA Flex Library Prep Kit. DNA yield will be determined fluorometrically using the High Sensitivity dsDNA kit on the Qubit® Fluorometer.
Biochemical and structural characterization of selected SAA end products by Western blot and solid-state NMR analysis | 12 months
  To study if SAA reaction products acquire biochemical (Western blot, densitometric quantitation), and structural (two-dimensional NMR spectra) characteristics useful to discriminate sALS, bALS and FTD or different phenotypes of the same disease. It is known that there is a clinical and neuropathological heterogeneity among these diseases. Through in-depth analyses of the SAA reaction products it will be possible to evaluate whether these differences are useful to obtain patient stratification.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Università degli Studi di Napoli "Federico II", Napoli
  - Azienda Ospedaliero Universitaria di Sassari, Sassari
  - Consorzio Interuniversitario Risonanze Magnetiche Metallo Proteine (CIRMMP), Sesto Fiorentino

IPD SHARING:
Plan to Share IPD: Yes
e-CRF created with RedCap
Supporting Information: ICF